CLINICAL TRIAL: NCT04437615
Title: Evaluation of the Clinical Performance of an Investigational Real-Time Colorectal Polyp Clinical Decision Support Device (CDSD)
Brief Title: Colorectal Polyp Clinical Decision Support Device Study
Acronym: CDSD
Status: Completed | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OCA 2019-GI-03
Record Dates: First submitted 2020-06-10; First posted 2020-06-18 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Polyp; Colorectal; Colonoscopy
Keywords: Colon; Polyp; Colorectal; Colonoscopy; AI; Narrow Band Imaging; Polyp Prediction; Artificial Intelligence
MeSH Terms: conditions — Polyps | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: The study shall be a prospective, single arm, multicenter study.
Masking Description: The pathologist (outcomes assessor) is blinded to the endoscopist predictions and CDSD prediction.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Single-arm (Experimental): CDSD un-aided vs. CDSD-aided predictions of diminutive polyp histology relative to ground-truth pathology. All patients will have both unaided and aided predictions.
  Interventions: Procedure: Colonoscopy; Device: Clinical Decision Support Device

INTERVENTIONS:
Procedure: Colonoscopy — Standard of care colonoscopy, with added use of CDSD as an adjunctive tool
Device: Clinical Decision Support Device — The investigational device consists of software residing on a dedicated computer enabling display of predicted diminutive polyp histology during colonoscopy.
  Other Names: CDSD

SUMMARY:
The study objective is to establish the efficacy of the colorectal polyp Clinical Decision Support Device (CDSD) in clinical use.

DETAILED DESCRIPTION:
Prospective, single arm, multicenter study with participating endoscopists comprising a range of clinical experience.

Consecutive consented patients meeting the entrance criteria will undergo standard colonoscopy with the adjunctive use of CDSD. Sensitivity and specificity of CDSD-unaided and CDSD-aided predictions will be compared with the ground truth of histopathology.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Willing and able to provide informed consent
* Subjects undergoing colonoscopy

Exclusion Criteria:

* Polyposis syndromes including Familial Adenomatous Polyposis Syndrome
* Inflammatory Bowel Disease
* Hereditary Non Polyposis Colorectal Cancer
* Severe coagulopathy
* Subjects scoring less than 6 on the Boston Bowel Prep Score or scoring less than 2 in any colon segment.
* No diminutive polyps detected during colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2379 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Borland Groover, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Immediately - 3 years

REFERENCES:
- [Derived] Rex DK, Bhavsar-Burke I, Buckles D, Burton J, Cartee A, Comar K, Edwards A, Fennimore B, Fischer M, Gerich M, Gilmore A, Hamdeh S, Hoffman J, Ibach M, Jackson M, James-Stevenson T, Kaltenbach T, Kaplan J, Kapur S, Kohm D, Kriss M, Kundumadam S, Kyanam Kabir Baig KR, Menard-Katcher P, Kraft C, Langworthy J, Misra B, Molloy E, Munoz JC, Norvell J, Nowak T, Obaitan I, Patel S, Patel M, Peter S, Reid BM, Rogers N, Ross J, Ryan J, Sagi S, Saito A, Samo S, Sarkis F, Scott FI, Siwiec R, Sullivan S, Wieland A, Zhang J, Repici A, Hassan C, Byrne MF, Rastogi A. Artificial Intelligence for Real-Time Prediction of the Histology of Colorectal Polyps by General Endoscopists. Ann Intern Med. 2024 Jul;177(7):911-918. doi: 10.7326/M24-0086. Epub 2024 May 21. PMID 38768450

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-arm
Started | 2379
Completed | 1290
Not Completed | 1089
Not completed — Screen Fails/Withdrawal | 1089

BASELINE CHARACTERISTICS:
Population: Eligible patients that rec'd a colonoscope and a successful CDSD prediction.
Arm/Group | Single-arm
Number analyzed (Participants) | 1252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 763
  >=65 years | 489
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 601
  Male | 651
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — During the screening process, patients were asked their race and ethnicity.
  Participants
    Caucasian | 976
    Asian | 19
    African American | 180
    Hispanic | 52
    Native American | 4
    Pacific Islander | 0
    Middle Eastern | 5
    Other | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1252

OUTCOME MEASURES:

1. Primary Outcome: Specificity and Sensitivity CDSD-unaided and CDSD-aided Endoscopist Predictions of Diminutive Polyp Histology
Description: CDSD-unaided and CDSD-aided predictions will be compared with the ground truth pathology results.
Time Frame: Upon receipt of pathology results (within one week)
Population: Total number of polyps from eligible participants (N=1252) who completed the study and had a successful CDSD prediction.
Measure: Number (95% Confidence Interval); unit: percentage of polyps
Units Other Than Participants: Number of polyps
Groups:
- CDSD Un-aided vs. CDSD-aided Predictions of Diminutive Polyp: CDSD un-aided vs. CDSD-aided predictions of diminutive polyp histology relative to ground-truth pathology. All patients will have both unaided and aided predictions.
  Colonoscopy: Standard of care colonoscopy, with added use of CDSD as an adjunctive tool
  Clinical Decision Support Device: The investigational device consists of software residing on a dedicated computer enabling display of predicted diminutive polyp histology during colonoscopy.
Arm/Group | CDSD Un-aided vs. CDSD-aided Predictions of Diminutive Polyp
Number analyzed (Participants) | 1252
Number analyzed (Number of polyps) | 2695
percentage of polyps
  Sensitivity for CDSD aided | 90.8 [89.3 to 92.3]
  Sensitivity for CDSD unaided | 90.7 [89.2 to 92.2]
  specificity for CDSD aided | 64.7 [61.7 to 67.8]
  specificity for CDSD unaided | 59.5 [56.6 to 62.7]

2. Secondary Outcome: 1. Number of Unaided NBI Prediction and Pathology Result of Diminutive Polyps Detected by the Endoscopist and Confirmed by Pathology for Which CDSD Does Not Return a Prediction.
Description: pathology as ground truth
Time Frame: Upon receipt of pathology results (within one week)
Population: Patients that completed the study.
Measure: Number; unit: number of polyps without CDSD prediction
Units Other Than Participants: Number of polyps
Groups:
- All Patients Who Completed the Study: All patients who completed the study and had NBI prediction
Arm/Group | All Patients Who Completed the Study
Number analyzed (Participants) | 1290
Number analyzed (Number of polyps) | 2807
number of polyps without CDSD prediction | 112

3. Secondary Outcome: 2. Sensitivity, Specificity, Negative Predictive Value (NPV), Positive Predictive Value (PPV) of Unaided Endoscopist Prediction Using White Light.
Description: pathology as ground truth
Time Frame: Upon receipt of pathology results (within one week)
Population: patients with polyps
Measure: Number; unit: percentage of polyps
Units Other Than Participants: number of Polyps
Groups:
- Unaided WLE Prediction Compared With Pathology: WLE prediction compared to pathology results
Arm/Group | Unaided WLE Prediction Compared With Pathology
Number analyzed (Participants) | 1252
Number analyzed (number of Polyps) | 2695
percentage of polyps
  Sensitivity | 88.5
  Specificity | 61.1
  Negative predictive value (NPV) | 74.7
  Positive predictive value (PPV) | 80.4

4. Secondary Outcome: 3. Sensitivity, Specificity, NPV, PPV of Unaided Endoscopist Prediction Using NBI Compared With Pathology.
Description: pathology as ground truth
Time Frame: Upon receipt of pathology results (within one week)
Population: Patients with polyps with NBI prediction
Measure: Number; unit: percentage of polyps
Units Other Than Participants: Number of Polyps
Groups:
- Unaided NBI Prediction Compared With Pathology: NBI prediction compared to pathology results
Arm/Group | Unaided NBI Prediction Compared With Pathology
Number analyzed (Participants) | 1252
Number analyzed (Number of Polyps) | 2695
percentage of polyps
  Sensitivity | 90.7
  Specificity | 59.5
  PPV | 74.6
  NPV | 83.8

5. Secondary Outcome: 4. Sensitivity, Specificity, NPV, PPV of CDSD Prediction Compared With Pathology.
Description: pathology as ground truth
Time Frame: Upon receipt of pathology results (within one week)
Population: Patients with CDSD prediction
Measure: Number; unit: percentage of polyps
Units Other Than Participants: Number of polyps
Groups:
- CDSD Prediction Compared With Pathology: CDSD prediction compared to pathology results
Arm/Group | CDSD Prediction Compared With Pathology
Number analyzed (Participants) | 1252
Number analyzed (Number of polyps) | 2695
percentage of polyps
  Sensitivity | 86.5
  Specificity | 69.5
  PPV | 78.6
  NPV | 79.9

6. Secondary Outcome: 5. Sensitivity, Specificity, NPV, PPV of CDSD-aided Endoscopist Prediction Compared With Pathology.
Description: pathology as ground truth
Time Frame: Upon receipt of pathology results (within one week)
Population: Aided CDSD prediction
Measure: Number; unit: percentage of polyps
Units Other Than Participants: Number of polyps
Groups:
- CDSD-Aided Prediction Compared With Pathology: Aided CDSD prediction compared to pathology results
Arm/Group | CDSD-Aided Prediction Compared With Pathology
Number analyzed (Participants) | 1252
Number analyzed (Number of polyps) | 2695
percentage of polyps
  Sensitivity | 90.8
  Specificity | 64.7
  PPV | 76.8
  NPV | 85.0

7. Secondary Outcome: 6. Number of Pathology Results for Diminutive Polyps With Discordant Unaided Predictions Using NBI and Aided Predictions With CDSD
Description: pathology as ground truth
Time Frame: Upon receipt of pathology results (within one week)
Population: NBI unaided prediction vs aided CDSD prediction
Measure: Number; unit: Polyps
Units Other Than Participants: Number of Polyps
Groups:
- Unaided Predictions Using NBI and Aided Predictions With CDSD Pathology: Unaided predictions using NBI and aided predictions with CDSD.
Arm/Group | Unaided Predictions Using NBI and Aided Predictions With CDSD Pathology
Number analyzed (Participants) | 1252
Number analyzed (Number of Polyps) | 2695
Polyps | 251

ADVERSE EVENTS:
Description: Deaths and adverse events were not collected.
Arm/Group | Single-arm
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT04437615/Prot_SAP_000.pdf